CLINICAL TRIAL: NCT04278300
Title: Study of the Discriminating Power of a Blood Biomarker for Omega-3 Polyunsaturated Fatty Acid Content of the Retina for Age-related Macular Degeneration (AMD)
Acronym: FATTY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CREUZOT 2019
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: patient with age-related exudative macular degeneration
  Interventions: Biological: blood sampling; Biological: faecal sampling (optional)
- control: Patient with no macular disorder and in need of cataract surgery
  Interventions: Biological: blood sampling; Biological: faecal sampling (optional)

INTERVENTIONS:
Biological: blood sampling — dosage of omega 3 polyunsaturated fatty acids, search for age-related macular degeneration susceptibility genese
Biological: faecal sampling (optional) — analysis of the microbiota by DNA sequencing

SUMMARY:
Age-related macular degeneration is a chronic degenerative retinal disease, which can lead to a progressive loss of visual acuity without affecting peripheral vision. It is a public health problem as it remains the leading cause of visual impairment in people over 50 years of age in industrialized countries.

Age-related macular degeneration has two clinical forms:

* Atrophic or dry form: progressive disappearance of photoreceptors, alteration of the pigmentary epithelium leading to a thinning of the macula.
* Exudative or humid form: development of immature choroidal neo-vessels, leading to the formation of edema or intra or sub-retinal hemorrhage at the origin of the symptoms.

There are still many questions about the pathogenesis of age-related macular degeneration, and there is currently no etiological treatment. The disorder is thought to have a multifactorial, genetic and environmental origin.

Among the environmental risk factors, dietary intake of omega-3 polyunsaturated acids and its effect on the retina are factors that influence both the incidence and progression of the disease. However, intervention studies have not been able to demonstrate the preventive value of omega-3 polyunsaturated fatty acids. It is likely that the precise identification of patients who could benefit from this supplementation is necessary. Currently, the estimation of dietary intake of omega-3 polyunsaturated fatty acids is based on dietary surveys, which implies a number of limits. A blood biomarker of omega-3 polyunsaturated fatty acid content in the retina has been previously identified, which if lowered may be a risk factor for age-related macular degeneration. A low level could also help to identify patients who would best respond to supplementation. A publication has been submitted and a patent has been filed for this biomarker. The objective of this project is to confirm the relationship between this biomarker and the presence of age-related macular degeneration. The analysis will be refined by correlating the discriminating character of the biomarker with factors that may influence the intestinal metabolism of dietary lipids and their bioavailability in the blood. For this purpose, the status of the subjects with regard to their intestinal flora (microbiota) will be evaluated. The relationship between lipid metabolism, microbiota and age-related macular degeneration should also provide a better understanding of the pathophysiological mechanisms that link diet, lipid metabolism and age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has provided written informed consent for participation in the study and genetic analyses
* Subject aged 50 years or older
* Subject with exudative AMD or
* Subject with macular disorder requiring cataract surgery

Exclusion Criteria:

* Person not affiliated to the national health insurance system
* Protected adults (curatorship, guardianship)
* Persons deprived of their liberty by judicial or administrative decision
* Adult unable to express consent
* Subject who has already participated in the study
* Subject with pre-existing maculopathy not labelled AMD
* Subject refusing blood sample
* Subject with diabetes
* Subject on antibiotics or having had an antibiotic treatment in the last 3 months
* Subject with a BMI < 18.5 or > 30 kg/m2
* Subject with extreme eating habits (veganism, bulimia, anorexia)
* Subject currently on a diet with avoidance of certain types of food or a low-calorie diet
* Subject with an inflammatory disease (especially digestive disease)
* Subject having undergone bariatric surgery
* Subject having digestive tract malformations

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients coming for consultation in the ophthalmology department
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Retinal Omega-3 polyunsaturated fatty acid levels | at inclusion

SECONDARY OUTCOMES:
Intestinal bacterial population levels | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France